CLINICAL TRIAL: NCT02655523
Title: A Comparison of Dexamethasone and Triamcinolone in Combination With Bupivacaine for Ultrasound-guided Occipital C2 Nerve Blocks: A Randomized Controlled Trial
Brief Title: A Comparison of Dexamethasone and Triamcinolone for Ultrasound-guided Occipital C2 Nerve Blocks
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00200460
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Triamcinolone; Triamcinolone Acetonide; Dexamethasone; Calcium Dobesilate; Saline Solution; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bupivacaine+Triamcinolone (Active Comparator): An ultrasound-guided C2 nerve block with 2 mL of 0.5% bupivacaine plus 1 mL 40 mg of triamcinolone.
  Interventions: Drug: Triamcinolone; Drug: Bupivacaine
- Bupivacaine+Dexamethasone (Active Comparator): An ultrasound-guided C2 nerve block with 2 mL of 0.5% bupivacaine plus 1 mL 4 mg of dexamethasone.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Bupivacaine+Saline (Placebo Comparator): An ultrasound-guided C2 nerve block with 2 mL of 0.5% bupivacaine plus 1 mL of preservative free normal saline.
  Interventions: Drug: Normal Saline; Drug: Bupivacaine

INTERVENTIONS:
Drug: Triamcinolone — 1 mL of 40 mg of Triamcinolone
  Other Names: Kenalog
  Arms: Bupivacaine+Triamcinolone
Drug: Dexamethasone — 1 mL of 4mg of Dexamethasone
  Other Names: Decadron
  Arms: Bupivacaine+Dexamethasone
Drug: Normal Saline — 1 mL of preservative free normal saline
  Other Names: 0.9% sodium chloride
  Arms: Bupivacaine+Saline
Drug: Bupivacaine — 2 mL of 0.5% bupivacaine
  Other Names: Sensorcaine

SUMMARY:
Greater occipital nerve (GON) injection is a commonly performed diagnostic and therapeutic procedure in headache patients. GON blocks have been shown to be effective in the treatment of a variety of headaches including occipital neuralgia, migraine, vascular headache, cluster headache, cervicogenic headache, and post-concussive headache. Local anesthetic and steroids have been successfully used for diagnostic and or therapeutic nerve pain such as lumbar radicultis with great success. Dexamethasone is a water soluble steroid, when combined with local anesthetic; it may increase the analgesia of block duration relative to its pharmacokinetics. When compared to dexamethasone, triamcinolone, a particulate steroid has a slower onset time but may provide anti-inflammatory effects up to several weeks. Investigators want to investigate to see if there exists a difference in reported pain intensity using the particulate anti-inflammatory corticosteroid (triamcinolone with bupivacaine) which may provide a greater reduction in reported pain intensity relief may allow the patient to undergo fewer interventional procedures.

DETAILED DESCRIPTION:
Greater occipital nerve (GON) injection is a commonly performed diagnostic and therapeutic procedure in headache patients. GON blocks have been shown to be effective in the treatment of a variety of headaches including occipital neuralgia, migraine, vascular headache, cluster headache, cervicogenic headache, and post-concussive headache.The GON provides sensory innervation to the posterior scalp to the vertex of the skull and is known to communicate with the third occipital nerve and lesser occipital nerve during its ascent at the occiput.The use of ultrasound guidance to assist with needle placement is becoming increasingly popular due to real-time visualization of soft tissue and surrounding vasculature as well as the appearance of bony structures. This imaging tool allows for fine adjustment of the needle tip and direct observation of the injectate thereby confirming local anesthetic spread at the targeted area. Local anesthetic and steroids have been successfully used for diagnostic and or therapeutic nerve pain such as lumbar radicultis with great success. Dexamethasone is a water soluble steroid, when combined with local anesthetic; it may increase the analgesia of block duration relative to its pharmacokinetics. When compared to dexamethasone, triamcinolone, a particulate steroid has a slower onset time but may provide anti-inflammatory effects up to several weeks. Investigators want to investigate to see if there exists a difference in reported pain intensity using the particulate anti-inflammatory corticosteroid (triamcinolone with bupivacaine) which may provide a greater reduction in reported pain intensity relief may allow the patient to undergo fewer interventional procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients, ≥ 18 years of age and under 75 years of age, presenting to the Northwestern Pain Center with occipital headaches who are scheduled to receive a ultrasound-guided occipital nerve block will be eligible for the study.
* Extracranial tenderness or Tinel's sign over the occipital nerve
* Poor response to other medical treatments (narcotics, physical therapy)
* Paroxysmal stabbing pain, with or without persistent aching between paroxysms, in the distribution(s) of the greater, lesser and/or third occipital nerves
* Visual Analog Scale (VAS) score of at least 4 at recent headache occurrence.

Exclusion Criteria:

* Abnormal cranial anatomy
* use of anticoagulants
* local infection
* refusal of or lack of consent
* pregnant patients
* systemic steroid in the last three months, steroid injection of any type in the last three months
* inability to read
* untreated/inadequately treated psychiatric disorders
* cannot comprehend or complete the questionnaires
* known allergies to local or steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
PROMIS (Patient Reported Outcome Measurement Information System) Pain Intensity Questionnaire | 2 weeks interval for up to 12 weeks
  Area under the PROMIS Pain Intensity Questionnaire T-score versus time profile for the 12 week study period

SECONDARY OUTCOMES:
Patients Global Impression of Change (PIGC) questionnaire | 2 week interval for for up to 12 weeks
  The Patient Global Impression of Change (PGIC) is a 7-point scale depicting a patient's rating of overall improvement.
Headache Under-Response to Treatment (HURT) questionnaire | Baseline and 3 month
  The HURT Questionnaire consists of eight questions which the patient answers as a measure of effectiveness of intervention against headache.

CONTACTS AND LOCATIONS:
Overall Officials: Antoun Nader, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Feingberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No